CLINICAL TRIAL: NCT06768944
Title: The Role of the Subjective Experience in Supporting Positive Effects Following Psilocybin: a Randomized, Controlled Clinical Trial Using Risperidone in Healthy Adults
Brief Title: Subjective Experience Following Psilocybin
Acronym: SEP-1
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Other
Other Study IDs: REB24-1121
Record Dates: First submitted 2024-12-16; First posted 2025-01-10 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Investigating the Importance of the Subjective Psychedelic Experience
Keywords: psychedelics; psilocybin; stress response; cortisol; healthy participants; risperidone; subjective effects
MeSH Terms: conditions — Fractures, Stress | interventions — Psilocybin; Risperidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- High-dose psilocybin + placebo (Active Comparator): placebo + 25 mg psilocybin (+60 min)
  Interventions: Drug: Psilocybin 25 mg; Drug: Placebo
- Low-dose psilocybin + placebo (Placebo Comparator): placebo + 1 mg psilocybin (+60 min)
  Interventions: Drug: Psilocybin 1 mg; Drug: Placebo
- High-dose psilocybin + risperidone (Experimental): 1 mg risperidone + 25 mg psilocybin (+60 min)
  Interventions: Drug: Psilocybin 25 mg; Drug: Risperidone 1 MG
- Low-dose psilocybin + risperidone (Active Comparator): 1 mg risperidone + 1 mg psilocybin (+60 min)
  Interventions: Drug: Psilocybin 1 mg; Drug: Risperidone 1 MG

INTERVENTIONS:
Drug: Psilocybin 25 mg — The drug product (DP) PEX010 is a capsule for oral administration and is manufactured with DS PYEX (12.5-14.0% psilocybin), excipients, and HPMC capsules. The product is manufactured in two product strengths, and this represents the high-dose (25mg)
  Other Names: PEX010; high-dose psilocybin
  Arms: High-dose psilocybin + placebo; High-dose psilocybin + risperidone
Drug: Psilocybin 1 mg — The drug product (DP) PEX010 is a capsule for oral administration and is manufactured with DS PYEX (12.5-14.0% psilocybin), excipients, and HPMC capsules. The product is manufactured in two product strengths, and this represents the low-dose (1mg)
  Other Names: PEX010; low-dose psilocybin
  Arms: Low-dose psilocybin + placebo; Low-dose psilocybin + risperidone
Drug: Risperidone 1 MG — risperidone 1mg capsules
  Other Names: Risperdal
  Arms: High-dose psilocybin + risperidone; Low-dose psilocybin + risperidone
Drug: Placebo — inactive placebo
  Arms: High-dose psilocybin + placebo; Low-dose psilocybin + placebo

SUMMARY:
The purpose of this study is to determine the importance of the acute subjective experience induced by psilocybin (the primary component of "magic mushrooms") in facilitating positive outcomes. Participants in this study will be given psilocybin in combination with either a placebo or risperidone, an atypical antipsychotic that block the subjective effects of psilocybin.

DETAILED DESCRIPTION:
The overall goal of this clinical trial is to systematically explore the relationship between the subjective psychedelic experience, improvements in well-being, and the stress response following psilocybin administration.

The investigators aim to determine whether blocking the acute subjective effects (via risperidone) will influence the acute or protracted effects of psilocybin as measured via self-report, biochemical, or psychophysiological measures. The study also aims to determine if individual variability in stress reactivity or regulation predicts acute (day of dosing) or protracted (1-week later) effects of psilocybin.

A single site will recruit 128 participants aged 18 to 65 who do not meet criteria for any psychiatric diagnoses. A series of questionnaires, blood labs, and medical exams including electrocardiogram will determine inclusion into the study. Once accepted into the study, participants will complete baseline measures assessing cortisol and brain-derived neurotrophic factor (BDNF) levels, cognitive flexibility, mood, well-being, personality traits, and anxiety levels.

Participants will then be randomly assigned into one of the following groups:

i) high dose psilocybin (25mg; "active dose") in combination with placebo pretreatment ii) high dose psilocybin (25mg; "active dose") in combination with risperidone pretreatment (1mg) iii) low dose psilocybin (1mg "active control") in combination with placebo pretreatment, iv) low dose psilocybin (1mg "active control") in combination with risperidone pretreatment (1mg).

Outcome measures will be assessed at 1-week and 1-month after each dosing session.

ELIGIBILITY:
Inclusion Criteria:

* Individuals of all sexes, gender identities, and ethnicities
* Ages 18 to 65 years of age at the time of screening
* Ability to read/write in English
* Agree not to consume psychoactive drugs 24 hours before dosing sessions or consume psychedelics during duration of study participation
* At least one self-reported positive experience prior to study participation with a psychoactive substance, specifically those known for altering perception or inducing hallucinatory effects (cannabis or psychedelics, including psilocybin, LSD, DMT, mescaline) or experience with non-pharmacological altered states of consciousness (meditation, breathwork)

Exclusion Criteria:

* Any notable abnormality on electrocardiogram or routine medical blood or urinalysis laboratory tests: I.e., unstable cardiac, renal, or liver disease, uncontrolled hypertension or diabetes, or other medical condition, as determined by the study staff, that could compromise participant safety
* Serious electrocardiogram abnormality, i.e., evidence of ischemia, myocardial infarction, QTc (Fridericia formula) prolongation (QTc > 0.45 for men, QTc > 0.47 for women).
* Abnormal liver enzymes (AST, ALT, GGT ≥4 times upper normal limit)
* Pre-existing low white blood cell count or a history of drug-induced leukopenia/neutropenia
* Insulin-dependent diabetes; if taking oral hypoglycemic agent, then no history of hypoglycemia
* History of epilepsy or seizures, neuroleptic malignant syndrome or tardive dyskinesia
* Hypertension (>140mmHg systolic or 90mmHg) or Tachycardia (HR >100bpm) as measures by best result of maximum of three vital sign recordings in a supine position after a 5 min resting period. Participants with a blood pressure not higher than 165/95 or a heart rate of not higher than 110bpm can be conditionally enrolled but dosing will only happen if the vitals at the dosing sessions are in the limits outlined above for inclusion.
* Current psychiatric diagnoses, such as major depressive disorder, generalized anxiety disorder, panic disorder, social anxiety disorder, obsessive compulsive disorder, moderate to severe substance use disorders, eating disorders, personality disorders, post-traumatic stress disorder
* Lifetime or current psychiatric diagnoses of psychosis, schizophrenia, bipolar disorder
* Family history: a first- or second degree relative with a history of schizophrenia or other psychotic disorders, bipolar I or II
* Medication: Any medication with the potential to interact with the investigational medicinal products, especially those with serotonergic mechanisms of actions like SSRIs, SNRIs or MAO-Inhibitors as well as other antipsychotics. Medication with potential drug-drug interactions (especially uridine 5'-diphospho-glucuronosyltransferase (UGT) and ALDH inhibitors and alcohol dehydrogenase (ADH) inhibitors for psilocybin and CYP2D6- and to a lesser extend CYP3A4 modulators for risperidone) are prohibited for at least 5 half-lives of the active moiety before the dosing.
* Serotonergic psychedelic use in the past 3 months (e.g. psilocybin, LSD, DMT, mescaline)
* Serious adverse events following previous psychedelic use
* Currently pregnancy or nursing, trying to become pregnant, or unwilling to use acceptable method of contraception during the study
* Acceptable methods of contraception include oral contraceptives, barrier with spermicide, IUD, medroxyprogesterone acetate (Depo Provera), contraceptive patch, vaginal contraceptive ring, or being post-menopausal or deemed medically unable to become pregnant (i.e., due to hysterectomy)
* Current or recent (within 12 weeks) participation in a clinical trial involving medication administration
* Any sensitivity or adverse reaction to previous use of a hallucinogen or risperidone
* Cognitive impairment (Folsetin Mini Mental State Exam score < 24)
* A disorder that may interfere with drug absorption, distribution, metabolism, or excretion (including gastrointestinal surgery).
* Suffered a traumatic brain injury with one of the following symptoms
* Loss of consciousness >30min
* Alteration of consciousness/mental state >24h
* Post-traumatic amnesia >1 day
* Glasgow Coma Scale (best available score in first 24 hours) <13
* The participant experienced a significant life event (such as pending loss of housing, family status change, loss of a close friend or relative) that could affect stability in the past 30 days.
* Any other circumstances that, in the opinion of the investigators, compromises participant safety

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Positive effects | One week and one month post-dosing
  Persisting Effects Questionnaire (PEQ) - 145 questions rated using a 6-point Likert scale from 0 to 6. There are 12 sub-scale themes assessing positive and negative changes in Attitudes About Life, Attitudes About Self, Mood Changes, Social Effects, Behavioural Changes, and Spirituality. Higher scores in the positive sub-scales indicate a better outcome, while higher scores in the negative sub-scales indicate a worse outcome.

SECONDARY OUTCOMES:
Stress reactivity | From start of dosing session to end of dosing session
  Stress reactivity will be assessed through heart rate variability
Biomarkers of stress and plasticity | from baseline to dosing session (one week post-baseline) to follow-up 1 (one week post doing session) to follow-up 2 (one month post dosing session)
  cortisol, ACTH, BDNF
Mood | from baseline to one week and one month post-dosing
  Mood will be assessed using the Positive and Negative Affect Schedule. The questionnaire has two sub-scales: the positive affect score (scores range from 10-50, higher scores represent better outcome) and the negative affect score (scores range from 10-50, higher scores represent worse outcome)
Well-being | from baseline to one week and one month post-dosing
  Well-being will be assessed using the Warwick-Edinburgh Mental Wellbeing Scale. The total score ranges from 14-70; a higher score represents a better outcome.
Anxiety | from baseline to one week and one month post-dosing
  Anxiety will be measured using the State-Trait Anxiety Inventory. The total score ranges from 20-80; a higher score represents a worse outcome.
Cognitive Flexibility | from baseline to one week and one month post-dosing
  The Berg Card Sorting Task is a set-shifting measure of cognitive flexibility modeled after the Wisconsin Card Sorting task. Participants must select the stimulus that is different from others based on feedback and adapt their responses once the criteria for correct choice switches. Perseverative errors are defined as the number of instances in which three incorrect responses are made based on a previous rule, and they are thought to reflect less cognitive flexibility (or cognitive rigidity).
Spontaneous Thought | from baseline to one week and one month post-dosing
  To measure spontaneous thought, participants will complete a Think Aloud task where they narrate their stream of thought in real time.
Reinforcement Learning | from baseline to one week and one month post-dosing
  Reinforcement learning will be assessed using a three-armed bandit task. This is a decision-making task in which participants must choose between three alternative targets whose values (probability of reward) changes over the trials.

CONTACTS AND LOCATIONS:
Overall Officials: Leah Mayo, PhD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No